CLINICAL TRIAL: NCT03893721
Title: Effect of Chronic Arsenic Exposure on Malnutrition Among Under-five Children Attending Assiut University Children Hospital
Brief Title: Effect of Chronic Arsenic Exposure on Malnutrition of Under Five Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, alyaa abdelaal mohamed abdelaal, principle investigator, Assiut University
Other Study IDs: 17100702
Record Dates: First submitted 2019-03-22; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Malnutrition, Child; Arsenic Poisoning Chronic
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Hair samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- malnourished under five children: children from 2 to 5 years with malnutrition
  Interventions: Diagnostic Test: arsenic exposure
- well nourished under five children: children from 2 to 5 years without malnutrition
  Interventions: Diagnostic Test: arsenic exposure

INTERVENTIONS:
Diagnostic Test: arsenic exposure — analysis of hair samples for Arsenic using Agilent graphite tube atomizer 120

SUMMARY:
Early life malnutrition is associated with later life health problems, Particularly Stunting, which is a height-for-age Z score less than -2 standard deviation of World Health Organization median.Underweight is weight-for-age Z score less than -2 standard deviation of World Health Organization median. Wasting is weight -for- height Z score less than -2 standard deviation of World Health Organization median.

DETAILED DESCRIPTION:
prevalence of under-five stunting, wasting and underweight are 21% and , 8% and 6% respectively in Egyptian Demographic Health Survey 2014.

The main risk factors for growth restriction in children are maternal under nutrition during pregnancy, lack of exclusive breastfeeding, inappropriate complementary feeding and micronutrient intake and high prevalence of enteric infections. However, other environmental exposures may also play a role in growth restriction .

High concentrations of Arsenic, lead and cadmium in placenta are associated with poor fetal out come and low birth weight. Arsenic crosses the placenta causing suppression of insulin-Like Growth Factor 1.

When breastfeeding is exclusive, infants are unlikely to be exposed to Arsenic by other routes of exposure such as external foods, drinking water and foods made at home using Arsenic contaminated water.

Rational of the study. Improvement of under-five nutritional status is a global target. Although the exposure to arsenic has increased globally, it's impact on nutritional status has seldom been investigated.

ELIGIBILITY:
Inclusion Criteria:

female children from 2 to 5 years

Exclusion Criteria:

Severely ill children other than severely malnourished.

* Children with congenital anomaly.
* Relatives.

Ages: 2 Years to 5 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Study Population: under five children attending Assiut university Children Hospital
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Chronic Arsenic Exposure of Under Five Children | one year
  Hair samples collected from participating children will be analyzed for Arsenic using Agilent graphite tube atomizer (GTA) 120
weight measurement | one year
  weight in kilograms will be measured to all participating children
height measurement | one year
  height in meters will be measured to all participating children

CONTACTS AND LOCATIONS:
Overall Officials: Alyaa Abdelaal, demonstrator, Principal Investigator — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Walker SP, Wachs TD, Gardner JM, Lozoff B, Wasserman GA, Pollitt E, Carter JA; International Child Development Steering Group. Child development: risk factors for adverse outcomes in developing countries. Lancet. 2007 Jan 13;369(9556):145-57. doi: 10.1016/S0140-6736(07)60076-2. PMID 17223478
- [Background] Milton AH, Attia J, Alauddin M, McEvoy M, McElduff P, Hussain S, Akhter A, Akter S, Islam MM, Ahmed AMS, Iyengar V, Islam MR. Assessment of Nutritional Status of Infants Living in Arsenic-Contaminated Areas in Bangladesh and Its Association with Arsenic Exposure. Int J Environ Res Public Health. 2018 Jan 2;15(1):57. doi: 10.3390/ijerph15010057. PMID 29301293
- [Background] Claus Henn B, Ettinger AS, Hopkins MR, Jim R, Amarasiriwardena C, Christiani DC, Coull BA, Bellinger DC, Wright RO. Prenatal Arsenic Exposure and Birth Outcomes among a Population Residing near a Mining-Related Superfund Site. Environ Health Perspect. 2016 Aug;124(8):1308-15. doi: 10.1289/ehp.1510070. Epub 2016 Feb 9. PMID 26859631
- [Background] Islam MR, Attia J, Alauddin M, McEvoy M, McElduff P, Slater C, Islam MM, Akhter A, d'Este C, Peel R, Akter S, Smith W, Begg S, Milton AH. Availability of arsenic in human milk in women and its correlation with arsenic in urine of breastfed children living in arsenic contaminated areas in Bangladesh. Environ Health. 2014 Dec 4;13:101. doi: 10.1186/1476-069X-13-101. PMID 25471535
- [Background] Vahter M. Health effects of early life exposure to arsenic. Basic Clin Pharmacol Toxicol. 2008 Feb;102(2):204-11. doi: 10.1111/j.1742-7843.2007.00168.x. PMID 18226075
- [Background] Signes-Pastor AJ, Cottingham KL, Carey M, Sayarath V, Palys T, Meharg AA, Folt CL, Karagas MR. Infants' dietary arsenic exposure during transition to solid food. Sci Rep. 2018 May 8;8(1):7114. doi: 10.1038/s41598-018-25372-1. PMID 29739998
- [Background] El-Badry AE-MA, Khalifa MM. Geochemical Assessment of Pollution at Manzala Lake, Egypt: Special Mention to Environmental and Health Effects of Arsenic, Selenium, Tin and Antimony. J Appl Sci [Internet]. 2017;17(2):72-80. Available from: http://dx.doi.org/10.3923/jas.2017.72.80
- [Background] El-Badry AE-MA, Khalifa MM. The occurrence and distribution of high-arsenic, selenium, tin and antimony in bottom sediments of Burullus lagoon and its effects on human health, Egypt. J African Earth Sci [Internet]. 2017 Dec 1 [cited 2019 Feb 23];136:305-11. Available from: https://www.sciencedirect.com/science/article/pii/S1464343X17303175?via%3Dihub